CLINICAL TRIAL: NCT05702411
Title: Air Stacking Technique For Pulmonary Reexpansion In The Ventilator After Expiratory Pause During Aspiration In Closed System
Brief Title: Air Stacking Technique For Pulmonary Reexpansion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 50845721.0.0000.5530
Record Dates: First submitted 2022-12-01; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Critical Care
Keywords: pulmonary reexpansion; air stacking; mechanical ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol 1 (Experimental): Closed system aspiration with an expiratory pause of 10 seconds followed by hyper insufflation maneuver with the Air Stacking technique.
  Interventions: Other: Air Stacking Technique
- Protocol 2 (Experimental): Closed system aspiration with an expiratory pause of 10 seconds.
  Interventions: Other: No Air Stacking Technique

INTERVENTIONS:
Other: Air Stacking Technique — Air Stacking lung reexpansion technique after aspiration with expiratory pause in a closed system.
  Arms: Protocol 1
Other: No Air Stacking Technique — Aspiration technique in a closed system of aspiration with an expiratory pause of 10 seconds.
  Arms: Protocol 2

SUMMARY:
A cross-over randomized clinical trial carried out at the Intensive Care Unit. Patients who are on mechanical ventilation for more than 24 hours will be included in the study. The following techniques will be applied: aspiration in a closed system with an expiratory pause of 10 seconds associated to hyperinflation maneuver with a mechanical ventilator with the Air Stacking technique and aspiration technique in a closed system of aspiration with an expiratory pause of 10 seconds.

DETAILED DESCRIPTION:
After randomization, all patients will be positioned in dorsal decubitus with the head elevated at 30 degrees and will be aspirated once with a closed suction system and with a vacuum limited to 150 cmH2O.

Two hours later, hemodynamic and ventilatory parameters will be collected and recorded.

If randomized to Protocol 1 (Air Stacking technique), the aspiration technique with closed system and expiratory pause will be performed three times during a 30-second interval, with a probe of the same caliber and the same vacuum value. One ml of saline solution will be instilled in the aspiration system to washing the closed suction circuit.

Immediately after, the Air Stacking maneuvers will be performed. If Protocol 2 (No Air Stacking technique), only tracheal suction with closed system.

Hemodynamic and ventilatory parameters will be collected after 1, 10 and 30 minutes of application. The secretions aspirated into the collection flasks will then be weighed, on a precision balance, by a collaborator blinded that is not part of the study, and the weight will be transcribed to the data collect.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years or older
* patients on mechanical ventilation for more than 48 hours
* patients on volume or pressure controlled ventilatory mode
* patients hemodynamically stable (equal mean blood pressure or more than 60 mmHg, and dose of Norepinephrine less than 1μg / Kg / minute)
* patients whose legal representatives authorize participation in the study.

Exclusion Criteria:

* undrained pneumothorax and hemothorax, and emphysema subcutaneous
* fracture of ribs
* ventilatory parameters with peak pressure greater than 40 cm/H2O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Tidal Volume (VT) (ml) | At 30-minute after the application of the studied technique.
  The tidal volume will be visualized directly at mechanical ventilation monitor. Variations in tidal volume will be considered before and after the interventions.

SECONDARY OUTCOMES:
Weight of secretion aspirated (grams) | Immediately after the application of one of the protocols.
  The secretion aspirated into the collection flask will be weighed on a precision laboratory scale.
Peripheral arterial oxygen saturation (SpO2) (%) | 1, 10 and 30-minute after the application of the studied technique.
  The SpO2 will be visualized on the monitor of the patient, and the value will be noted.
Peak inspiratory pressure (PIP) (cm H2O) | 1, 10 and 30-minute after the application of the studied technique.
  The PIP will be visualized directly at mechanical ventilation monitor, and the value will be noted.
End expiratory pressure (PEEP) (cmH2O) | 1, 10 and 30-minute after the application of the studied technique.
  The PEEP will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Air trapping (AUTO-PEEP) (cmH2O) | 1, 10 and 30-minute after the application of the studied technique.
  The AUTO-PEEP will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Mechanical ventilation circuit pressure (cmH2O) | 1, 10 and 30-minute after the application of the studied technique.
  The mechanical ventilation circuit pressure will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Endotracheal tube diameter (ETT) (mm) | 1-minute after the application of the studied technique.
  The endotracheal tube diameter is directly written in the product package.
Dynamic compliance (Cd) (ml/cmH2O) | 1, 10 and 30-minute after the application of the studied technique.
  The Cd will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Resistance (R) (L/s) | 1, 10 and 30-minute after the application of the studied technique.
  The R will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Drive pressure (cmH2O) | 1, 10 and 30-minute after the application of the studied technique.
  The drive pressure will be calculated by the difference between plateau pressure and positive end-expiratory pressure in the mechanical ventilation, and the value will be noted.
Heart rate (HR) (beats per minute) | 1, 10 and 30-minute after the application of the studied technique.
  The HR will be visualized on the monitor of the patient, and the value will be noted.
Respiratory rate (RR) (breaths per minute) | 1, 10 and 30-minute after the application of the studied technique.
  The RR will be visualized on the monitor of the patient, and the value will be noted.
Mean arterial pressure (MAP) (mmHg) | 1, 10 and 30-minute after the application of the studied technique.
  The MAP will be calculated using the systolic and diastolic blood pressure, and the value will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda M Kutchak, Master, Principal Investigator — Grupo Hospitalar Conceição
Locations (1):
- Hospital Cristo Redentor, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slutsky AS. History of Mechanical Ventilation. From Vesalius to Ventilator-induced Lung Injury. Am J Respir Crit Care Med. 2015 May 15;191(10):1106-15. doi: 10.1164/rccm.201503-0421PP. PMID 25844759
- [Background] Walter JM, Corbridge TC, Singer BD. Invasive Mechanical Ventilation. South Med J. 2018 Dec;111(12):746-753. doi: 10.14423/SMJ.0000000000000905. PMID 30512128
- [Background] Pham T, Brochard LJ, Slutsky AS. Mechanical Ventilation: State of the Art. Mayo Clin Proc. 2017 Sep;92(9):1382-1400. doi: 10.1016/j.mayocp.2017.05.004. PMID 28870355
- [Background] Van der Schans CP. Bronchial mucus transport. Respir Care. 2007 Sep;52(9):1150-6; discussion 1156-8. PMID 17716383
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Niel-Weise BS, Snoeren RL, van den Broek PJ. Policies for endotracheal suctioning of patients receiving mechanical ventilation: a systematic review of randomized controlled trials. Infect Control Hosp Epidemiol. 2007 May;28(5):531-6. doi: 10.1086/513726. Epub 2007 Mar 22. PMID 17464911
- [Background] Ciesla ND. Chest physical therapy for patients in the intensive care unit. Phys Ther. 1996 Jun;76(6):609-25. doi: 10.1093/ptj/76.6.609. PMID 8650276
- [Background] Branson RD. Secretion management in the mechanically ventilated patient. Respir Care. 2007 Oct;52(10):1328-42; discussion 1342-7. PMID 17894902
- [Background] American Association for Respiratory Care. AARC Clinical Practice Guidelines. Endotracheal suctioning of mechanically ventilated patients with artificial airways 2010. Respir Care. 2010 Jun;55(6):758-64. PMID 20507660
- [Background] Pagotto IM, Oliveira LR, Araujo FC, Carvalho NA, Chiavone P. Comparison between open and closed suction systems: a systematic review. Rev Bras Ter Intensiva. 2008 Dec;20(4):331-8. English, Portuguese. PMID 25307236
- [Background] Lopes FM, Lopez MF. Impact of the open and closed tracheal suctioning system on the incidence of mechanical ventilation associated pneumonia: literature review. Rev Bras Ter Intensiva. 2009 Mar;21(1):80-8. English, Portuguese. PMID 25303133
- [Background] de Fraga Gomes Martins L, da Silva Naue W, Skueresky AS, Bianchi T, Dias AS, Forgiarini LA. Effects of Combined Tracheal Suctioning and Expiratory Pause: A Crossover Randomized Clinical Trial. Indian J Crit Care Med. 2019 Oct;23(10):454-457. doi: 10.5005/jp-journals-10071-23263. PMID 31749553
- [Background] Stiller K. Physiotherapy in intensive care: an updated systematic review. Chest. 2013 Sep;144(3):825-847. doi: 10.1378/chest.12-2930. PMID 23722822
- [Background] Smith DJ, Gaffney EA, Blake JR. Modelling mucociliary clearance. Respir Physiol Neurobiol. 2008 Nov 30;163(1-3):178-88. doi: 10.1016/j.resp.2008.03.006. Epub 2008 Mar 20. PMID 18439882
- [Background] Karamaoun C, Sobac B, Mauroy B, Van Muylem A, Haut B. New insights into the mechanisms controlling the bronchial mucus balance. PLoS One. 2018 Jun 22;13(6):e0199319. doi: 10.1371/journal.pone.0199319. eCollection 2018. PMID 29933368
- [Background] Pieterse A, Hanekom SD. Criteria for enhancing mucus transport: a systematic scoping review. Multidiscip Respir Med. 2018 Jul 6;13:22. doi: 10.1186/s40248-018-0127-6. eCollection 2018. PMID 29988934
- [Background] Konrad F, Schiener R, Marx T, Georgieff M. Ultrastructure and mucociliary transport of bronchial respiratory epithelium in intubated patients. Intensive Care Med. 1995 Jun;21(6):482-9. doi: 10.1007/BF01706201. PMID 7560491
- [Background] Savian C, Paratz J, Davies A. Comparison of the effectiveness of manual and ventilator hyperinflation at different levels of positive end-expiratory pressure in artificially ventilated and intubated intensive care patients. Heart Lung. 2006 Sep-Oct;35(5):334-41. doi: 10.1016/j.hrtlng.2006.02.003. PMID 16963365
- [Background] Coppadoro A, Bellani G, Foti G. Non-Pharmacological Interventions to Prevent Ventilator-Associated Pneumonia: A Literature Review. Respir Care. 2019 Dec;64(12):1586-1595. doi: 10.4187/respcare.07127. Epub 2019 Sep 24. PMID 31551284
- [Background] AGÊNCIA NACIONAL DE VIGILÂNCIA SANITÁRIA. Medidas de Prevenção de Infecção Relacionada à Assistência à Saúde.; 2017.
- [Background] Franca EE, Ferrari F, Fernandes P, Cavalcanti R, Duarte A, Martinez BP, Aquim EE, Damasceno MC. Physical therapy in critically ill adult patients: recommendations from the Brazilian Association of Intensive Care Medicine Department of Physical Therapy. Rev Bras Ter Intensiva. 2012 Mar;24(1):6-22. English, Portuguese. PMID 23917708
- [Background] Naue Wda S, da Silva AC, Guntzel AM, Condessa RL, de Oliveira RP, Rios Vieira SR. Increasing pressure support does not enhance secretion clearance if applied during manual chest wall vibration in intubated patients: a randomised trial. J Physiother. 2011;57(1):21-6. doi: 10.1016/S1836-9553(11)70003-0. PMID 21402326
- [Background] van der Schans CP, Postma DS, Koeter GH, Rubin BK. Physiotherapy and bronchial mucus transport. Eur Respir J. 1999 Jun;13(6):1477-86. doi: 10.1183/09031936.99.13614879. PMID 10445628
- [Background] Ardehali SH, Fatemi A, Rezaei SF, Forouzanfar MM, Zolghadr Z. The Effects of Open and Closed Suction Methods on Occurrence of Ventilator Associated Pneumonia; a Comparative Study. Arch Acad Emerg Med. 2020 Jan 11;8(1):e8. eCollection 2020. PMID 32021989
- [Background] Letchford E, Bench S. Ventilator-associated pneumonia and suction: a review of the literature. Br J Nurs. 2018 Jan 11;27(1):13-18. doi: 10.12968/bjon.2018.27.1.13. PMID 29323990
- [Background] Taggart JA, Dorinsky NL, Sheahan JS. Airway pressures during closed system suctioning. Heart Lung. 1988 Sep;17(5):536-42. PMID 3417464
- [Background] Palazzo SG, Soni B. Pressure changes during tracheal suctioning--a laboratory study. Anaesthesia. 2013 Jun;68(6):576-84. doi: 10.1111/anae.12218. PMID 23662749
- [Background] Santos FR, Schneider Junior LC, Forgiarini Junior LA, Veronezi J. Effects of manual rib-cage compression versus PEEP-ZEEP maneuver on respiratory system compliance and oxygenation in patients receiving mechanical ventilation. Rev Bras Ter Intensiva. 2009 Jun;21(2):155-61. English, Portuguese. PMID 25303345
- [Background] Spapen HD, De Regt J, Honore PM. Chest physiotherapy in mechanically ventilated patients without pneumonia-a narrative review. J Thorac Dis. 2017 Jan;9(1):E44-E49. doi: 10.21037/jtd.2017.01.32. PMID 28203436
- [Background] Rosa FK, Roese CA, Savi A, Dias AS, Monteiro MB. [Behavior of the lung mechanics after the application of protocol of chest physiotherapy and aspiration tracheal in patients with invasive mechanical ventilation]. Rev Bras Ter Intensiva. 2007 Jun;19(2):170-5. Portuguese. PMID 25310775
- [Background] Jones A, Rowe BH. Bronchopulmonary hygiene physical therapy in bronchiectasis and chronic obstructive pulmonary disease: a systematic review. Heart Lung. 2000 Mar-Apr;29(2):125-35. PMID 10739489
- [Background] Hodgson C, Denehy L, Ntoumenopoulos G, Santamaria J, Carroll S. An investigation of the early effects of manual lung hyperinflation in critically ill patients. Anaesth Intensive Care. 2000 Jun;28(3):255-61. doi: 10.1177/0310057X0002800302. PMID 10853205
- [Background] Unoki T, Kawasaki Y, Mizutani T, Fujino Y, Yanagisawa Y, Ishimatsu S, Tamura F, Toyooka H. Effects of expiratory rib-cage compression on oxygenation, ventilation, and airway-secretion removal in patients receiving mechanical ventilation. Respir Care. 2005 Nov;50(11):1430-7. PMID 16253149
- [Background] Avena Kde M, Duarte AC, Cravo SL, Sologuren MJ, Gastaldi AC. [Effects of manually assisted coughing on respiratory mechanics in patients requiring full ventilatory support]. J Bras Pneumol. 2008 Jun;34(6):380-6. doi: 10.1590/s1806-37132008000600008. Portuguese. PMID 18622505
- [Background] Brito MF, Moreira GA, Pradella-Hallinan M, Tufik S. Air stacking and chest compression increase peak cough flow in patients with Duchenne muscular dystrophy. J Bras Pneumol. 2009 Oct;35(10):973-9. doi: 10.1590/s1806-37132009001000005. English, Portuguese. PMID 19918629
- [Background] Iskandar K, Sunartini, Nugrahanto AP, Ilma N, Kalim AS, Adistyawan G, Siswanto, Naning R. Use of air stacking to improve pulmonary function in Indonesian Duchenne muscular dystrophy patients: bridging the standard of care gap in low middle income country setting. BMC Proc. 2019 Dec 16;13(Suppl 11):21. doi: 10.1186/s12919-019-0179-4. eCollection 2019. PMID 31890014
- [Background] Pattanshetty RB, Gaude GS. Effect of multimodality chest physiotherapy in prevention of ventilator-associated pneumonia: A randomized clinical trial. Indian J Crit Care Med. 2010 Apr;14(2):70-6. doi: 10.4103/0972-5229.68218. PMID 20859490
- [Background] Pattanshetty RB, Gaude GS. Effect of multimodality chest physiotherapy on the rate of recovery and prevention of complications in patients with mechanical ventilation: a prospective study in medical and surgical intensive care units. Indian J Med Sci. 2011 May;65(5):175-85. PMID 23364504
- [Background] Pepe PE, Marini JJ. Occult positive end-expiratory pressure in mechanically ventilated patients with airflow obstruction: the auto-PEEP effect. Am Rev Respir Dis. 1982 Jul;126(1):166-70. doi: 10.1164/arrd.1982.126.1.166. PMID 7046541
- [Background] Natalini G, Tuzzo D, Rosano A, Testa M, Grazioli M, Pennestri V, Amodeo G, Marsilia PF, Tinnirello A, Berruto F, Fiorillo M, Filippini M, Peratoner A, Minelli C, Bernardini A; VENTILAB Group. Assessment of Factors Related to Auto-PEEP. Respir Care. 2016 Feb;61(2):134-41. doi: 10.4187/respcare.04063. Epub 2015 Nov 24. PMID 26604329
- [Background] Bugedo G, Retamal J, Bruhn A. Does the use of high PEEP levels prevent ventilator-induced lung injury? Rev Bras Ter Intensiva. 2017 Apr-Jun;29(2):231-237. doi: 10.5935/0103-507X.20170032. PMID 28977263
- [Background] Volpe MS, Adams AB, Amato MB, Marini JJ. Ventilation patterns influence airway secretion movement. Respir Care. 2008 Oct;53(10):1287-94. PMID 18811989
- [Background] Fink JB. Forced expiratory technique, directed cough, and autogenic drainage. Respir Care. 2007 Sep;52(9):1210-21; discussion 1221-3. PMID 17716387
- [Background] Lasocki S, Lu Q, Sartorius A, Fouillat D, Remerand F, Rouby JJ. Open and closed-circuit endotracheal suctioning in acute lung injury: efficiency and effects on gas exchange. Anesthesiology. 2006 Jan;104(1):39-47. doi: 10.1097/00000542-200601000-00008. PMID 16394688
- [Background] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Background] Das A, Cole O, Chikhani M, Wang W, Ali T, Haque M, Bates DG, Hardman JG. Evaluation of lung recruitment maneuvers in acute respiratory distress syndrome using computer simulation. Crit Care. 2015 Jan 12;19(1):8. doi: 10.1186/s13054-014-0723-6. PMID 25578295
- [Background] Goligher EC, Hodgson CL, Adhikari NKJ, Meade MO, Wunsch H, Uleryk E, Gajic O, Amato MPB, Ferguson ND, Rubenfeld GD, Fan E. Lung Recruitment Maneuvers for Adult Patients with Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S304-S311. doi: 10.1513/AnnalsATS.201704-340OT. PMID 29043837
- [Background] Hartland BL, Newell TJ, Damico N. Alveolar recruitment maneuvers under general anesthesia: a systematic review of the literature. Respir Care. 2015 Apr;60(4):609-20. doi: 10.4187/respcare.03488. Epub 2014 Nov 25. PMID 25425708
- [Background] Corley A, Sharpe N, Caruana LR, Spooner AJ, Fraser JF. Lung volume changes during cleaning of closed endotracheal suction catheters: a randomized crossover study using electrical impedance tomography. Respir Care. 2014 Apr;59(4):497-503. doi: 10.4187/respcare.02601. Epub 2013 Sep 17. PMID 24046466
- [Background] Almgren B, Wickerts CJ, Hogman M. Post-suction recruitment manoeuvre restores lung function in healthy, anaesthetized pigs. Anaesth Intensive Care. 2004 Jun;32(3):339-45. doi: 10.1177/0310057X0403200306. PMID 15264727
- [Background] Chicayban LM. Acute effects of ventilator hyperinflation with increased inspiratory time on respiratory mechanics: randomized crossover clinical trial. Rev Bras Ter Intensiva. 2019 Oct 14;31(3):289-295. doi: 10.5935/0103-507X.20190052. eCollection 2019. PMID 31618346
- [Background] Rothen HU, Neumann P, Berglund JE, Valtysson J, Magnusson A, Hedenstierna G. Dynamics of re-expansion of atelectasis during general anaesthesia. Br J Anaesth. 1999 Apr;82(4):551-6. doi: 10.1093/bja/82.4.551. PMID 10472221
- [Background] Dohna-Schwake C, Ragette R, Teschler H, Voit T, Mellies U. IPPB-assisted coughing in neuromuscular disorders. Pediatr Pulmonol. 2006 Jun;41(6):551-7. doi: 10.1002/ppul.20406. PMID 16617451
- [Background] Toussaint M, Pernet K, Steens M, Haan J, Sheers N. Cough Augmentation in Subjects With Duchenne Muscular Dystrophy: Comparison of Air Stacking via a Resuscitator Bag Versus Mechanical Ventilation. Respir Care. 2016 Jan;61(1):61-7. doi: 10.4187/respcare.04033. Epub 2015 Oct 6. PMID 26443018
- [Background] Maggiore SM, Lellouche F, Pigeot J, Taille S, Deye N, Durrmeyer X, Richard JC, Mancebo J, Lemaire F, Brochard L. Prevention of endotracheal suctioning-induced alveolar derecruitment in acute lung injury. Am J Respir Crit Care Med. 2003 May 1;167(9):1215-24. doi: 10.1164/rccm.200203-195OC. Epub 2003 Feb 13. PMID 12615633